CLINICAL TRIAL: NCT04782726
Title: Radiation Therapy Plan Quality Improvement Using Ideal Theoretical Isodose Distribution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 20-0114; HSC20200678H (Other: UT Health Science Center San Antonio IRB)
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Placebo Comparator): After consent and study enrollment the subject will be scheduled for CT simulation for radiation treatment planning. At the time of CT simulation, they will be immobilized by means of a thermoplastic mask. For patients in the control arm, the radiation treatment planning will proceed as normal. Treatment planning is performed on Pinnacle. The patient will return for validation of the radiation plan. Validation involves collecting on-table X-rays or cone beam CTs when the patient is in position for treatment, which is the standard of care. Most often, the date of validation will happen within 5 business days of the CT simulation.
  Interventions: Other: Radiation therapy
- Research Arm (Experimental): After consent and study enrollment the subject will be scheduled for CT simulation for radiation treatment planning. At the time of CT simulation, they will be immobilized by means of a thermoplastic mask. For patients in the research arm, a theoretical plan will be created after physician's segmentation and will be used as a guide for the final plan. The patient will return for validation of the radiation plan. Validation involves collecting on-table X-rays or cone beam CTs when the patient is in position for treatment, which is the standard of care. Most often, the date of validation will happen within 5 business days of the CT simulation.
  Interventions: Other: Software Solution for Radiation Therapy Treatment; Other: Radiation therapy

INTERVENTIONS:
Other: Software Solution for Radiation Therapy Treatment — Software has been developed for individualized pre optimization evaluation of the patient anatomy and prescribed dose of radiation therapy.
  Other Names: Treatment planning
  Arms: Research Arm
Other: Radiation therapy — Standard of Care planning for Radiation therapy is used to treat the subjects for head and neck cancer
  Other Names: Radiation treatment

SUMMARY:
The researchers hope that based on the study findings future patients may benefit from a more precise radiation treatment plan that can be developed more quickly and thus decrease the time from Computerized Tomography Simulation to start of treatment.

DETAILED DESCRIPTION:
As part of this study participants will receive the standard of care treatment for all head and neck cancer patients. The researchers plan to use a software program to see if it will assist in developing the best radiation treatment plan possible. The researchers will also measure the quality of each treatment plan so areas of improvement can be identified.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Ability to provide informed written consent in either English or Spanish.
* Patient planned to undergo radiation therapy for Head and Neck Cancer.

Exclusion Criteria:

* Current pregnancy, as this is a contraindication to receiving radiation therapy.
* History of prior radiotherapy to the head and neck.
* Any condition or history as evidenced by patient record and/or self-report that, in the opinion of the investigator, would interfere with adherence to daily radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Mean radiation dose to Organs at Risk (OAR) | Baseline to last treatment (up to 33 treatments or about 7 weeks)
  Measurement of radiation dose to organs at risk. The goal is to maintain the PTV (Planning Target Volume) coverage while minimizing the dose to organs at risk (OARs).
Maximum radiation dose to Organs at Risk (OAR) | Baseline to last treatment (up to 33 treatments or about 7 weeks)
  Measurement of maximum radiation dose to organs at risk. The goal is to maintain the PTV (Planning Target Volume) coverage while minimizing the dose to organs at risk (OARs).

SECONDARY OUTCOMES:
Time required to plan radiation therapy dose | CT Simulation to first treatment (about 1 week)
  The time required with and without individualized pre optimization information will be recorded and compared to determine efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios Stathakis, PhD, Principal Investigator — UT Health San Antonio
Locations (1):
- Mays Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No